CLINICAL TRIAL: NCT02444650
Title: Photoplethysmogram Measurement of Pulse Wave Velocity
Brief Title: Measurement of Pulse Wave Velocity
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: QATP2804
Record Dates: First submitted 2015-04-29; First posted 2015-05-14 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: Correlation; pulse wave velocity measurement; tonometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pulse wave velocity measurement Photoplethysmogram — Correlation of pulse wave velocity measurement.
Device: tonometer

SUMMARY:
Optically-based data will be compared to tonometry to determine correlation of pulse wave velocity measurement.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of18-25 and 65-90 will be studied.
* Normotensive and hypertensive subjects
* Willing to provide informed consent

Exclusion Criteria:

* has finger deformities or amputations that will prohibit proper sensor placement
* pregnant or actively trying to get pregnant
* Cardiogreen or other intravascular/tissue dyes less than 5 hours prior to the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy normotensive and hypertensive subjects.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Optically based pulse wave velocity measurement correlation to the tonometry measure. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Curry, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States